CLINICAL TRIAL: NCT00371254
Title: Phase II Study of Dasatinib (BMS-354825) for Advanced 'Triple-negative' Breast Cancer
Brief Title: A Study of Dasatinib (BMS-354825) in Patients With Advanced 'Triple-negative' Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Study Director, Bristol-Myers Squibb
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CA180-059
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Results first posted 2011-03-15 (Estimated); Last update posted 2011-03-15 (Estimated); Status verified 2011-02

CONDITIONS: Breast Cancer; Metastasis
Keywords: Recurrent, locally-advanced, or 'triple negative' metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Neoplasm Metastasis; Recurrence | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: Dasatinib
- 2 (Experimental)
  Interventions: Drug: Dasatinib

INTERVENTIONS:
Drug: Dasatinib — Tablets, Oral, 100 mg, twice daily as long as the patient benefits (avg <6 months)
  Other Names: Sprycel; BMS-354825
  Arms: 1
Drug: Dasatinib — Tablets, Oral, 70 mg, twice daily as long as the patient benefits (avg <6 months)
  Arms: 2

SUMMARY:
This study will determine whether the investigational drug dasatinib is effective in treatment of women with progressive advanced triple-negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* females, 18 or older
* recurrent or progressive locally advanced, or 'triple negative' metastatic breast cancer
* paraffin-embedded tissue block must be available
* measurable disease
* prior chemotherapy with an anthracycline, a taxane, or both (neoadjuvant, adjuvant, or metastatic setting)
* 0, 1 or 2 chemotherapies in the metastatic setting
* adequate organ function

Exclusion Criteria:

* Metastatic disease confined to bone only
* Symptomatic CNS metastasis
* Concurrent medical condition which may increase the risk of toxicity
* Unable to take oral medication

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2006-12; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (10):
- United States (5):
  - Ucsf-Comprehensive Cancer Center, San Francisco, California
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - Dana-Farber Cancer Inst, Boston, Massachusetts
  - Montefiore Medical Center, The Bronx, New York
  - University Of Texas Md Anderson Cancer Ctr, Houston, Texas
- France (2):
  - Local Institution, Paris
  - Local Institution, Toulouse
- Local Institution, Modena, Italy
- Spain (2):
  - Local Institution, Barcelona
  - Local Institution, Lleida

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 55 participants were enrolled in the study; 11 discontinued prior to study drug administration (8 no longer met study criteria, 2 other reasons and 1 administrative reason by the sponsor)
Groups:
- Dasatinib 100 mg BID: Participants were administered an oral dose of 100 mg dasatinib tablet twice daily for a total daily dose (TDD) of 200 mg. Study treatment continued for as long as it was tolerated, or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
- Dasatinib 70 mg BID: Participants were administered an oral dose of 70 mg dasatinib tablet twice daily for a TDD of 140 mg. Study treatment continued for as long as it was tolerated, or until PD, defined as appearance of new lesion/s, or >=20% increase in the sum of the LD of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Period: Overall Study
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Started | 23 (Number of participants treated) | 21 (Number of participants treated)
Completed | 0 (Number of participants remained on study till the study drug could be tolerated) | 0 (Number of participants remained on study till the study drug could be tolerated)
Not Completed | 23 | 21
Not completed — Disease progression | 13 | 13
Not completed — Study drug toxicity | 3 | 5
Not completed — Subject request | 5 | 0
Not completed — Investigator Decision | 2 | 0
Not completed — Adverse event unrelated to study drug | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID | Total
Number analyzed (Participants) | 23 | 21 | 44
Age, Customized [Number; unit: participants]
  <50 years | 4 | 9 | 13
  >=50 years | 19 | 12 | 31
Age Continuous [Mean (Standard Deviation); unit: years] | 56.4 (8.98) | 51.5 (9.34) | 54.0 (9.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 9 | 12 | 21
  Unknown or Not Reported | 11 | 7 | 18
Race/Ethnicity, Customized [Number; unit: participants]
  White | 20 | 19 | 39
  Black or African American | 2 | 1 | 3
  Asian | 0 | 1 | 1
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR)
Description: Tumor response was defined as the number of participants whose best response was CR or PR, per the Response Evaluation Criteria in Solid Tumor (RECIST): CR: disappearance of all target/non-target lesions; PR: >= 30% decrease in the sum of the LDs of target lesions relative to the baseline sum LD.
Time Frame: Baseline to end of study drug therapy (up to 65 weeks).
Population: All response-evaluable participants i.e. all treated participants who had at least 1 measurable lesion at baseline, had at least 1 on-study tumor assessment or discontinued before any on-study tumor assessment for reasons related to disease or study drug.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
participants | 2 | 0

2. Secondary Outcome: Number of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) at or After 16 Weeks on Study
Description: The number of participants whose best response was CR, PR or SD (per the RECIST) at or after 16 weeks on study: CR: disappearance of all target/non-target lesions; PR: >=30% decrease in the sum of the LDs of target lesions relative to baseline sum LD; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PD: appearance of new lesion/s, or >=20% increase in the sum of the LD of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to 16 weeks.
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
Participants | 3 | 1

3. Secondary Outcome: Percentage of Participants With Complete Response (CR), Partial Response (PR) or Stable Disease (SD) at or After 16 Weeks on Study
Description: The percentage of participants whose best response was CR, PR or SD (per the RECIST) at or after 16 weeks on study: CR: disappearance of all target/non-target lesions; PR: >=30% decrease in the sum of the LDs of target lesions relative to baseline sum LD; SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD; PD: appearance of new lesion/s, or >=20% increase in the sum of the LD of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Time Frame: Baseline to 16 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
percentage of participants | 13.04 [2.78 to 33.59] | 5.0 [0.13 to 24.87]

4. Secondary Outcome: Proportion of Participants With Progression-Free Survival (PFS) at Weeks 9, 17, and 25
Description: PFS:time from first dose until the date that progressive disease (PD) or clinical PD (cPD) observed,per RECIST criteria.PD:appearance of new lesion/s,or >=20% increase in the sum of the LD of target lesions,relative to smallest sum LD recorded since treatment start,or unequivocal progression of existing non-target lesions;cPD:deterioration related to disease requiring treatment discontinuation,but without radiographic PD.Participants who died without PD were considered to have PD on the date of death.For participants who neither progressed nor died,date of the last tumor assessment was used.
Time Frame: Weeks 9, 17, and 25
Population: All treated participants
Measure: Number; unit: Proportion of Participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
Proportion of Participants
  Week 9 | 0.40 (0.13) | 0.35 (0.12)
  Week 17 | 0.32 (0.13) | 0.14 (0.09)
  Week 25 | 0.21 (0.12) | 0.00 (0.00)

5. Secondary Outcome: Mean Number of Weeks of Complete Response (CR) or Partial Response (PR)
Description: Mean number of weeks of CR/PR (time from first date of CR/PR until first date PD observed. Tumor response defined per RECIST: CR: disappearance of all target/non-target lesions; PR: >=30% decrease in sum of LDs of target lesions relative to baseline sum LD; PD: appearance of new lesion or >=20% increase in sum of LD of target lesions relative to smallest sum LD or unequivocal progression of existing non-target lesions. Participants who died without reported PD were considered to have PD on date of death. For participants who neither progressed nor died, date of last tumor assessment used.
Time Frame: Baseline to end of study drug therapy (up to 53.86 weeks)
Population: Response-evaluable participants who achieved a complete response (CR) or partial response (PR)
Measure: Mean (Full Range); unit: weeks
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 2 | 0
weeks | 31 [8.14 to 53.86] |

6. Secondary Outcome: Mean Plasma Concentration at Week 3
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose and 1, 3, 6 and 12 hours after each dose administration
Population: Participants who were evaluable for pharmacokinetic analysis. "n" signifies the number of participants evaluable at each time point.
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Groups:
- Dasatinib 50 mg BID: Participants were administered an oral dose of 50 mg dasatinib tablet twice daily for a total daily dose (TDD) of 100 mg. Study treatment continued for as long as it was tolerated, or until progressive disease (PD), defined as appearance of new lesion/s, or >=20% increase in the sum of the longest diameter (LD) of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID | Dasatinib 50 mg BID
Number analyzed (Participants) | 10 | 10 | 1
nanograms (ng)/mL
  0 hour (n = 10, 10, 1) | 9.02 (3.79) | 7.14 (4.41) | 2.88 (NA) — Number of participants too small.
  1 hour (n = 10, 10, 1) | 103.35 (80.94) | 66.41 (47.53) | 35.05 (NA) — Number of participants too small.
  3 hour (n = 10, 10, 1) | 50.98 (35.23) | 35.47 (21.51) | 32.58 (NA) — Number of participants too small.
  6 hour (n = 10, 10, 1) | 19.02 (8.43) | 14.28 (8.78) | 10.35 (NA) — Number of participants too small.
  12 hour (n = 7, 6, 1) | 9.11 (3.39) | 15.43 (17.60) | 3.60 (NA) — Number of participants too small.

7. Primary Outcome: Percentage of Participants With Complete Response (CR) or Partial Response (PR)
Description: The percentage of participants whose best response was CR or PR, per the RECIST: CR: disappearance of all target/non-target lesions; PR: >= 30% decrease in the sum of the LDs of target lesions relative to the baseline sum LD.
Time Frame: Baseline to end of study drug therapy (up to 65 weeks).
Population: All response-evaluable participants i.e. all treated participants who had at least 1 measurable lesion at baseline, 1 on-study tumor assessment or discontinued before any on-study tumor assessment for reasons related to disease or study drug were included in this dataset.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
percentage of participants | 8.7 [1.07 to 28.04] | 0.0 [0.0 to 0.0]

8. Secondary Outcome: Mean Plasma Concentration at Week 7
Description: Mean plasma concentration was obtained directly from the concentration-time data.
Time Frame: At pre-dose and 1, 3, 6 and 12 hours after each dose administration
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: nanograms (ng)/mL
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 10 | 10
nanograms (ng)/mL
  0 hour (n = 2, 6) | 8.87 (0.49) | 4.89 (2.16)
  1 hour (n = 2, 6) | 120.92 (23.16) | 84.36 (62.01)
  3 hour (n = 3, 6) | 37.04 (2.26) | 44.80 (12.40)
  6 hour (n = 2, 6) | 15.75 (0.14) | 14.25 (4.69)
  12 hour (n = 1, 5) | 8.39 (NA) — Number of participants too small. | 18.87 (30.11)

9. Secondary Outcome: Mean Change in Concentration of Collagen Type IV From Baseline
Description: Collagen Type IV is a measure of anti-angiogenic activity. Plasma samples for assessment of change in concentration of Collagen Type IV were obtained and analyzed by enzyme-linked immunosorbent assay.
Time Frame: Baseline, Week 3 and Week 5
Population: Participants who were evaluable for pharmacodynamic analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: percentage of baseline
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
percentage of baseline
  Week 3 (n = 17, 12) | 39.51 [28.60 to 51.34] | 26.92 [12.06 to 43.76]
  Week 5 (n = 8, 11) | 34.31 [17.46 to 53.58] | 35.18 [15.80 to 57.82]

10. Secondary Outcome: Mean Change in Concentration of Vascular Endothelial Growth Factor Receptor-2 (VEGFR2) From Baseline
Description: VEGFR2 is a measure of anti-angiogenic activity. Plasma samples for assessment of change in concentration of VEGFR2 were obtained and analyzed by enzyme-linked immunosorbent assay.
Time Frame: Baseline, Week 3 and Week 5
Population: Participants who were evaluable for pharmacodynamic analysis.
Measure: Geometric Mean (90% Confidence Interval); unit: percentage of baseline
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 20
percentage of baseline
  Week 3 (n = 17, 12) | 25.07 [17.73 to 32.86] | 18.59 [13.12 to 24.32]
  Week 5 (n = 8, 11) | 33.56 [22.23 to 45.94] | 25.12 [17.59 to 33.12]

11. Secondary Outcome: Percentage Change in Tumor Biomarkers
Description: Tumor markers are indicators of tumor activity which may be used to predict clinical benefit and circulating biomarkers may reveal key mechanisms of action. Tissue staining was performed for caveolin, phospho-caveolin, EphA2 and insulin-like growth factor binding protein 2 (IGFBP2) markers using immunohistochemistry assays.
Time Frame: Baseline
Population: All treated participants who were evaluable for the analysis. These data for tumor markers were integrated with those from other studies and are not reportable for this study alone.
Measure: Median (Inter-Quartile Range); unit: percentage
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 0 | 0

12. Secondary Outcome: Profiling of Messenger-ribonucleic Acid (mRNA) Expression: mRNA Signal Intensity
Description: Pharmacogenomic analysis included the assessment of the relationship between clinical benefit and mRNA expression levels and between clinical benefit and protein phosphorylation. Tumor mRNA expression was analyzed in all available tissues. mRNA was extracted from 96 formalin-fixed paraffin-embedded tissue (FFPET) samples, amplified, and fluorescently labeled. Gene expression profiling was conducted using Affymetrix Human Genome U133A 2.0 DNA microarrays. mRNA expression is reported as quantile normalized RMA values.
Time Frame: Baseline
Population: All treated participants who were evaluable for the analysis. These data for pharmacogenomic analyses were integrated with those from other studies and are not reportable for this study alone.
Measure: Number; unit: log2 scale (unitless)
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 0 | 0

13. Secondary Outcome: Number of Participants Who Died, Experienced Other Serious Adverse Events (SAEs) or Adverse Events (AEs)
Description: An AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition (even if not caused by the study drug). An SAE was defined as an AE that resulted in death, was life-threatening, required hospitalization (or prolongation of existing hospitalization), or was an important medical event.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants.
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Death | 1 | 0
  Serious adverse events (SAEs) | 11 | 3
  All adverse events (AEs) | 23 | 21

14. Secondary Outcome: Number of Participants Who Experienced Drug-related SAEs, Drug-related AEs, Drug-related Grade 3 AEs and Discontinuations Due to Drug-related AEs
Description: AE=any new untoward medical occurrence/worsening of pre-existing medical condition.SAE=AE that resulted in death, was life-threatening, required hospitalization (or prolongation of existing hospitalization), or was an important medical event. Drug-related SAEs or AEs are those events with relationship to study therapy of certain, probable or possible.AEs were graded using the National Cancer Institute (NCI) Common Toxicity Criteria (CTC), v3: Grade 1=mild, 2=moderate, 3=severe, 4=life threatening, 5=death.Participants who discontinued the study due to any drug-related AEs were also recorded.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Drug-related SAEs | 5 | 1
  Drug-related AEs | 23 | 19
  Drug-related Grade 3 AEs | 12 | 8
  Drug-related AEs Leading to Discontinuation | 4 | 6

15. Secondary Outcome: Most Frequent Drug-related Adverse Events (AEs)
Description: Most frequent drug-related AEs are those AEs with frequency >=25% in either group. Drug-related AEs are those events with relationship to study therapy of certain, probable or possible.
Time Frame: From start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Diarrhea | 12 | 7
  Fatigue | 10 | 14
  Nausea | 10 | 14
  Dyspnea | 10 | 6
  Pleural Effusion | 9 | 7
  Rash | 9 | 5
  Headache | 8 | 4
  Anorexia | 9 | 0
  Vomiting | 7 | 6
  Cough | 7 | 5
  Abdominal pain | 7 | 0

16. Secondary Outcome: Number of Participants With Grade 3 or 4 Abnormalities in Hematology Measurements
Description: Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening. Grades 3 and 4 criteria are defined as follows: Granulocytes: Grade 3 <1.0 - 0.5 x 10^9/L; Grade 4, <0.5 x 10^9/L. Hemoglobin: Grade 3, <8.0 - 6.5 g/dL; Grade 4, <6.5 g/dL. Platelets: Grade 3, <50.0 - 25.0 x 10^9/L; Grade 4, <25.0 x 10^9/L. Leukocytes: Grade 3, <2.0 - 1.0 x 10^9/L; Grade 4, <1.0 x 10^9/L.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Granulocytes | 3 | 0
  Hemoglobin | 0 | 0
  Platelet Count | 0 | 0
  Leukocytes | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormalities (Grade 1 or 2) in Prothrombin Time (PT)
Description: PT is a measure of the clotting ability of the blood. Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening and 5=death.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Grade 1 | 3 | 0
  Grade 2 | 0 | 0

18. Secondary Outcome: Number of Participants With Abnormalities (Grade 1 or 2) in Partial Thromboplastin Time (PTT)
Description: PTT is a measure of the clotting ability of the blood. Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1=mild, Grade 2=moderate, Grade 3=severe, Grade 4=life-threatening and 5=death.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants.
Measure: Number; unit: Participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Grade 3 or 4 Serum Chemistry Abnormalities in Alanine Aminotransferase (ALT), Aspartate Aminotransferase (AST) and Alkaline Phosphatase
Description: Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening. Grade 3 and 4 criteria are defined as follows: ALT, AST and alkaline phosphatase: Grade 3: >5-20 x upper limit of normal (ULN), Grade 4: >20 x ULN.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Alkaline phosphatase | 1 | 1
  Alanine aminotransferase | 1 | 3
  Aspartate aminotransferase | 0 | 3

20. Secondary Outcome: Number of Participants With Grade 3 or 4 Serum Chemistry Abnormalities in Calcium, Potassium, Magnesium and Sodium
Description: Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening. Grade 3 and 4 criteria are defined as follows: Calcium: Grade 3-4 : <6.0 - <7.0 or >12.5 - >13.5 mg/dL, Potassium: Grade 3-4 : <2.5 - <3.0 or >6.0 - >7.0 mEq/L, Magnesium: Grade 3-4 : <0.6 - <0.8 or >2.46 - >6.6 mEq/L, Sodium:< 120- 130 or >155 - >160 mEq/L.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  High calcium | 0 | 0
  Low calcium | 0 | 1
  High potassium | 0 | 0
  Low potassium | 1 | 0
  High magnesium | 0 | 0
  Low magnesium | 0 | 0
  High sodium | 0 | 0
  Low sodium | 0 | 0

21. Secondary Outcome: Number of Participants With Grade 3 or 4 Serum Chemistry Abnormalities in Creatinine, Bicarbonate, Inorganic Phosphorous and Bilirubin (Total).
Description: Abnormalities were graded according to the NCI CTC, version 3.0: Grade 1 = mild, Grade 2 = moderate, Grade 3 = severe, Grade 4 = life threatening. Grade 3 and 4 criteria are defined as follows: Creatinine: Grade 3-4 : > 3.0 -6.0 ULN (upper limit of normal),Bicarbonate: Grade 3-4: <16 -<22 mEq/L, Phosphorous: Grade 3-4 : <1.0 - <2.0 mg/dL, Bilirubin, total: Grade 3-4: >3.0 - >10.0 ULN.
Time Frame: Throughout study, from start of study drug therapy up to 30 days after the last dose.
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants
  Creatinine | 0 | 0
  Bicarbonate | 0 | 0
  Inorganic Phosphorus | 1 | 2
  Bilirubin, Total | 0 | 0

22. Secondary Outcome: Number of Participants With Identified Electrocardiogram (ECG) Abnormalities
Description: ECGs were performed and all recordings were evaluated by the investigator. Abnormalities, if present at any study time point, were listed. The following ECG variables were collected: heart rate, PR interval, QRS width, and QT interval. Abnormalities in ECGs were defined by reference to institutional reports.
Time Frame: Baseline, Weeks 3, 9, 17 and 25, then every 8 weeks until the end of study treatment (up to 17 weeks).
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants | 4 | 3

23. Secondary Outcome: Number of Participants With Abnormal Vital Signs Measurements
Description: Vital signs included systolic and diastolic blood pressure and heart rate. The investigator used his or her judgement to decide whether or not the values were abnormal.
Time Frame: At each study visit (Week 3, 5, 7, 9, 13, 17 and 25) and end of treatment (up to 17 weeks)
Population: All treated participants
Measure: Number; unit: participants
Arm/Group | Dasatinib 100 mg BID | Dasatinib 70 mg BID
Number analyzed (Participants) | 23 | 21
participants | 0 | 0

ADVERSE EVENTS:
Groups:
- All Participants: All treated participants who were administered a twice-daily oral dose of either 100 mg (TDD 200 mg) or 70 mg (TDD 140 mg) dasatinib tablet. Study treatment continued for as long as it was tolerated, or until PD, defined as appearance of new lesion/s, or >=20% increase in the sum of the LD of target lesions, relative to the smallest sum LD recorded since treatment start, or unequivocal progression of existing non-target lesions.
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 14/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=44)
MYOPERICARDITIS (Cardiac disorders) | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 2
HYPOTENSION (Vascular disorders) | 2
NAUSEA (Gastrointestinal disorders) | 1
ASCITES (Gastrointestinal disorders) | 1
VOMITING (Gastrointestinal disorders) | 2
DYSPHAGIA (Gastrointestinal disorders) | 1
CONSTIPATION (Gastrointestinal disorders) | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 1
INFECTION (Infections and infestations) | 1
PNEUMONIA (Infections and infestations) | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 1
PERIORBITAL OEDEMA (Skin and subcutaneous tissue disorders) | 1
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1
COSTOCHONDRITIS (Musculoskeletal and connective tissue disorders) | 1
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 3
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1
PYREXIA (General disorders) | 2
GENERALISED OEDEMA (General disorders) | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 1
MALIGNANT NEOPLASM PROGRESSION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | All Participants (N=44)
DRY EYE (Eye disorders) | 3
WEIGHT DECREASED (Investigations) | 5
ALANINE AMINOTRANSFERASE (Investigations) | 4
ASPARTATE AMINOTRANSFERASE (Investigations) | 4
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 3
FLUSHING (Vascular disorders) | 4
HOT FLUSH (Vascular disorders) | 5
ANXIETY (Psychiatric disorders) | 5
INSOMNIA (Psychiatric disorders) | 7
HEADACHE (Nervous system disorders) | 15
DIZZINESS (Nervous system disorders) | 3
PARAESTHESIA (Nervous system disorders) | 3
NAUSEA (Gastrointestinal disorders) | 25
VOMITING (Gastrointestinal disorders) | 14
DIARRHOEA (Gastrointestinal disorders) | 20
DYSPEPSIA (Gastrointestinal disorders) | 3
STOMATITIS (Gastrointestinal disorders) | 4
CONSTIPATION (Gastrointestinal disorders) | 10
ABDOMINAL PAIN (Gastrointestinal disorders) | 8
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 4
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 3
URINARY TRACT INFECTION (Infections and infestations) | 3
ANOREXIA (Metabolism and nutrition disorders) | 12
ANAEMIA (Blood and lymphatic system disorders) | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 4
RASH (Skin and subcutaneous tissue disorders) | 16
ERYTHEMA (Skin and subcutaneous tissue disorders) | 3
PRURITUS (Skin and subcutaneous tissue disorders) | 4
MYALGIA (Musculoskeletal and connective tissue disorders) | 8
BACK PAIN (Musculoskeletal and connective tissue disorders) | 6
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 6
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 4
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 3
COUGH (Respiratory, thoracic and mediastinal disorders) | 17
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 19
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 15
PAIN (General disorders) | 3
FATIGUE (General disorders) | 25
PYREXIA (General disorders) | 7
ASTHENIA (General disorders) | 8
CHEST PAIN (General disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.